CLINICAL TRIAL: NCT00483587
Title: A Safety and Efficacy Study to Evaluate Intravenous Heme Arginate Infusion in Patients With an Acute Coronary Syndrome Without ST-elevation (NSTEMI)
Brief Title: Does Heme Oxygenase-1 Induction Ameliorate Cardiac Injury After Myocardial Infarction?
Acronym: HAEM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: W.T. Ruifrok, University Medical Centre Groningen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WTR-ECG-1; EudraCT 2006-006389-40
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Acute Myocardial Infarction
Keywords: NSTEMI; Acute coronary syndrome; Heme arginate; HO-1; Heme oxygenase-1
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome | interventions — heme arginate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Heme arginate — 1-3 x heme arginate infusion, in 30 minutes iv. Heme arginate is dissolved in 250 ml NACl.

SUMMARY:
Rationale: A safety and dose defining study in which the investigators hypothesize that in patients with acute coronary syndrome without ST-elevation (NSTEMI) treatment with heme arginate results in better clinical outcome by inducing the heme oxygenase-1 (HO-1) pathway.

Objective: 1) Is induction of HO-1 and its degradation products, especially bilirubin, safe in patients with an acute coronary syndrome without ST-elevation; 2) What is the optimal effective dose to administer in patients with NSTEMI; 3) Are HO-1 and its degradation products endogenously activated in patients with acute coronary syndrome; 4) Does treatment with heme arginate result in a less cardiac damage; 5) Which other cardioprotecting pathways are activated by administration of heme arginate?

Study population: Male and female patients with confirmed acute coronary syndrome without ST-elevation, between 18 - 80 yr old.

Intervention: 10 patients receive a single administration of heme arginate (3 mg/kg), administered intravenously in 15 minutes directly after admission; 10 patients receive two administrations of heme arginate (3 mg/kg) on day 0 and 1; 10 patients receive three administrations of heme arginate (3 mg/kg) on day 0, 1 and 2 after admission, administered intravenously in 15 minutes. To determine endogenous levels of HO-1 and time course of HO-1 activation after NSTEMI, blood is drawn and the same assays are performed in 15 patients with NSTEMI. As controls for the blood tests, blood is drawn and the same assays are performed in 15 patients with non-typical angina pectoris in whom no cardiac disease could be detected from the investigators out-patient clinic.

Main study parameters/endpoints: The primary endpoint is the incidence rate of adverse events between the three treated groups. This includes hemodynamic monitoring, rhythm monitoring and biochemical and hematological difference between the three treated groups. Secondary endpoints are the differences from baseline between heme arginate treated groups in activity of the HO-1 pathway, including, but not limited to, HO-1 activity, free heme, bilirubin (direct and indirect) levels, serum ferritin, and carbon monoxide (CO). Furthermore, differences between heme arginate treated groups on NTproBNP, CK-MB and Troponin T and difference between heme arginate treated subjects in LVEF measured by echocardiography, 3 and 7 days and 6 months after NSTEMI.

DETAILED DESCRIPTION:
The interventional part of this study is a single centre safety and dose defining pilot study in which patients are allocated to heme arginate infusion for 1 day (hem-1d), heme arginate infusion for 2 days, or heme arginate infusion during 3 days (hem-3d) in consecutive order. So, the three patient groups consist of three intervention groups.

Based upon the pharmacokinetic data in porphyria patients (3 mg/kg/day for 4-7 days), the investigators rationalize that 3 fixed doses of heme arginate will be the optimal dose to counter attack the acute phase after NSTEMI. Longer infusion of heme arginate seems at this moment not rational.

The investigators will first administer in 10 patients 1 dose of heme arginate (hem-1d, day 0) to assess safety. If safety is assured in the hem-1d group, 10 patients will receive two days of heme arginate infusion (day 0 and 1). After this group is completed and safety is assured, the third group (n = 10) will receive heme arginate infusion in three consecutive days after NSTEMI (day 0, 1 and 2 after admission).

Heme arginate is considered safe in NSTEMI patients if no adverse events occur in the consecutive groups. To assess safety during the course of the study the following possible events are monitored:

* New onset of myocardial infarction with ST-elevation (STEMI);
* Cardiac decompensation;
* Sustained ventricular arrhythmia requiring defibrillation;
* All cause death;
* Drop of mean arterial blood pressure (MAP) of more than 20 mmHg (MAP is defined as 2 x diastolic blood pressure + 1 x systolic blood pressure divided by 3 (MAP = 2 x Pdias + Psys / 3));
* Eosinophilia (> 0.5 x 109/l) in combination with fever and/or rash and/or shivering or anaphylactic shock;
* Renal insufficiency (serum creatinine above 300 µmol/l);
* ASAT or ALAT are elevated to at least 3 times the upper limit of normal;
* Severe hematological abnormalities, defined as thrombocytopenia < 40 x 109/l, leucocytopenia < 2.0 x 109/l, or hemolytic anemia;
* Activated partial thromboplastin time (aPTT) elevated to at least 3 times the upper limit of normal;
* Severe bleeding, defined as requiring blood transfusion.

In the event one of the above mentioned effects occur, the investigators will report this to the METC and deliberate before continuing the study. If, after deliberation with the METC, heme arginate turns out not to be safe in NSTEMI patients, the inclusion of patients will be terminated immediately and all patients who already received heme arginate will be followed thoroughly. The investigator will take care that all subjects are kept informed.

After completion of each group the METC will be informed about the progress of the study.

Regardless of allocation, all patients will receive care as usual according to national/international guidelines 79, 80.

Patients with NSTEMI, admitted to the University Medical Center Groningen (UMCG), are asked to participate in the study and will sign informed consent. After signing consent, blood is drawn via venipuncture for baseline data.

On day 0, 1, 2, 3, 7, and 180 after NSTEMI blood is drawn for additional measurements. Echocardiography is performed to determine left ventricular function, including left ventricular ejection fraction (LVEF), after 3 days, 7 days and 180 days. To assess the possible anti-hypertensive component of heme arginate treatment, 24 hour ambulatory blood pressure recordings will be conducted at day 7 and 6 months after NSTEMI.

The following components of the heme pathway will be determined: free heme, hemoglobin, ferritin, carbon monoxide, heme oxygenase (HO)-1, biliverdin, and direct and non direct bilirubin. To monitor safety, the investigators will evaluate liver enzymes (ALAT, ASAT, γ-GT, AP, LDH), clotting times (INR, APTT, PT), electrolytes (Na, K, Cl, Mg) and furthermore regular hematology (Hb, Ht, thrombocytes) and chemistry (Blood Urea Nitrogen, Creatinine, CK, CK-MB, Troponin T, Brain Natriuretic Peptide, VEGF and Erythropoietin).

All participants will also be asked for blood to assess DNA polymorphisms affecting HO-1 activity, such as HO-1 polymorphisms, and for assessment of quality of endothelial progenitor cells (EPCs).

Total number included patients into the interventional part of this study will be 30 patients. Follow-up is completed 6 months after inclusion of the last patient. The investigators estimate inclusion will take approximately 6 months. The study duration therefore comes to a total of at least 12 months. The maximal duration of the study will be 18 months, including analysis of the results.

In addition, two groups of patients will be asked in the non-interventional part of this study:

1. The investigators hypothesize that due to the acute coronary syndrome HO-1 is activated, but at too low levels to have clinical benefit. To determine the time course for HO-1 activity and its degradation products after NSTEMI, the investigators will draw blood and perform all the same assays in 15 patients with NSTEMI as described above. It is not possible to use the same assays executed in the interventional part of this study, for heme arginate infusion will interfere with the outcomes.
2. As healthy controls for the blood tests and to gain insight in normal levels of HO-1 activity, the investigators will draw blood and do the same baseline assays in 15 patients with non-typical angina pectoris in whom no cardiac disease could be detected from our out-patient clinic.

All these patients will be asked to participate in the non-intervention part of this study, receive a separate information letter and will sign an informed consent form. If consent is given, blood is drawn via venipuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for the interventional part of this study

   * Before any study-specific procedures, the appropriate written informed consent must be obtained.
   * Male and female between 18 to 80 years of age.
   * Having NSTEMI confirmed by elevated CK (CK-total (>200 U/l), CK-MB act, CK-mass (>5.00 µg/l) and/or Troponin T (>0.01µg/l) levels.
2. Inclusion criteria for the non-interventional part of this study

   * Before any study-specific procedures, the appropriate written informed consent must be obtained.
   * Male en female between 18 and 80 years of age.

     * 15 patients having NSTEMI confirmed by elevated CK (CK-total (>200 U/l), CK-MB act, CK-mass (>5.00 µg/l) and/or Troponin T (>0.01µg/l)levels.
     * 15 patients with non-typical angina pectoris in whom no cardiac disease could be detected.

Exclusion Criteria:

1. Exclusion criteria for the interventional part of this study

   * ST-elevation on the electrocardiogram.
   * An unstable medical condition, defined as having been hospitalized for a noncardiac condition within 4 weeks of screening, or otherwise unstable in the judgment of the investigator (e.g. at risk of complications or adverse events unrelated to study participation).
   * Younger than 18 and older than 80 years of age.
   * Normal levels of CK en Troponin T.
   * Clinical history of chronic kidney disease (at any point prior to registration).
   * Any known hepatic disease.
   * Recent (within 3 months) history of alcohol or illicit drug abuse disorder, based on self report.
   * Clinically significant abnormality in chemistry, hematology, or urinalysis parameters performed within the screening period.
   * Participation in any investigational device or drug trial(s) or receiving investigational agent(s) within 30 days.
   * Any condition (e.g. psychiatric illness, etc.) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
   * Legally incompetent adults, for which reason what so ever.
   * Any known hypersensitivity/allergic reaction to one of the constituents of heme arginate (hemin, L-arginin, propylene glycol, ethanol).
   * Any known hypersensitivity/allergic reaction to any known drugs or constituents of medication.
2. Exclusion criteria for the non-interventional part of this study

   * ST-elevation on the electrocardiogram.
   * An unstable medical condition, defined as having been hospitalized for a noncardiac condition within 4 weeks of screening, or otherwise unstable in the judgment of the investigator.
   * Younger than 18 and older than 80 years of age.
   * Clinical history of metabolic diseases, e.g. chronic kidney disease, hepatic disease or otherwise in the investigator's opinion.
   * Clinically significant abnormality in chemistry, hematology, or urinalysis parameters performed within the screening period.
   * Participation in any investigational device or drug trial(s) or receiving investigational agent(s) within 30 days.
   * Legally incompetent adults, for which reason what so ever.
   * For the 15 patients which act as controls for the NSTEMI patients: no history for cardiac disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Subject's incidence rates of adverse events between the three treated groups with heme arginate | 6 months
Difference between the three intervention groups in liver enzymes levels (ASAT, ALAT, γ-GT, AP, LDH), blood clotting factor parameters ((INR, APTT, PT) and electrolytes (Na, K, Cl, Mg)) as safety monitoring of heme arginate administration. | 6 months

SECONDARY OUTCOMES:
Difference from baseline between heme arginate treated groups in activity of the HO-1 pathway, including, but not limited to, HO-1 activity, free heme, bilirubin (direct and indirect) levels, serum ferritin, and CO. | 6 months
Difference between heme arginate treated groups on NTproBNP, CK-MB and Troponin T. | 6 months
Difference between heme arginate treated groups in LVEF measured by echocardiography, 3 and 7 days and 6 months after NSTEMI. | 6 months
The time course of HO-1 activation after NSTEMI, including, but not limited to, HO-1 activity, free heme, bilirubin (direct and indirect) levels, serum ferritin, and CO. | 6 months
Basal levels of HO-1 activity, including, but not limited to, free heme, bilirubin (direct and indirect) levels, serum ferritin, and CO. | 6 months
DNA polymorphisms affecting HO-1 activity. | 6 months
Which other cardioprotecting pathways are activated by administration of heme arginate (e.g. serum levels of erythropoietin, VEGF and number of circulating EPCs)? | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. F. Zijlstra, MD, PhD, Principal Investigator — University Medical Centre Groningen, Dept. of Cardiology
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands